CLINICAL TRIAL: NCT06752031
Title: Optimization of Care and Recovery in Older Colorectal Surgery Patients: A Hybrid Effectiveness-Implementation Pilot Study Protocol
Brief Title: Optimizing Care Transition Process for Older Colorectal Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sevdenur Cizginer Konuk, MD, MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K76AG078620-02 (NIH)
Record Dates: First submitted 2024-12-18; First posted 2024-12-30 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Surgery; Care Transition; Older Adults (65 Years and Older)
Keywords: Colorectal surgery; Care transition; Older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OSCAR-S Care Transition Model (Experimental): The surgery nurse coach within the OSCAR-S model will provide touch points to patients and families to support their transition from hospital to home after surgery.
  Interventions: Behavioral: OSCAR-S Care Transition Model

INTERVENTIONS:
Behavioral: OSCAR-S Care Transition Model — Patients and families in the intervention arm will receive touch points from the surgery nurse coach to support their care transition from hospital to home after surgery.

SUMMARY:
The goal of this study to test if a care transition intervention designed for older colorectal surgery patients would improve outcomes after discharge. It will assess the feasibility of the intervention.

DETAILED DESCRIPTION:
The period following discharge poses particularly high risks for older colorectal surgery patients. Nearly a quarter of these patients are readmitted within a month of discharge due to a variety of issues including medication errors, surgical complications, imbalance in fluid or nutrition, or worsening of pre-existing chronic diseases.Recognizing the complex interplay of these factors, it isa more comprehensive approach is imperative to improve post- operative patient care. Geriatrics co-management programs incorporate interdisciplinary patient management approaches and geriatric principles to improve outcomes in older surgical patients.The OSCAR program is an integrated care model developed by geriatricians in collaboration with colorectal surgeons that combines geriatrics co-management with postoperative surgical care for older colorectal surgery patients. The care transition intervention (CTI) is a well-established care transition model that focuses on four domains at discharge: 1) medication self-management, 2) the personal health record, 3) timely primary care/specialty care follow-up, and 4) knowledge of red flags that indicate a worsening in condition. CTI involves interactions with a trained transition coach, both in-person visits and phone calls over four weeks. In this study, the goal is to bridge the gap between inpatient and post-discharge phases and mitigate the risk of hospital readmissions through adaptation and combination of the core components of a geriatric surgery core co-management (OSCAR) program with the core components of a care transition (CTI) program by applying an implementation research approach. By customizing OSCAR co-management model with the CTI intervention model, the investigators will leverage their strengths and, efficiently address the unique requirements of both patients and the healthcare environment. The investigators will conduct a pilot feasibility hybrid type I implementation effectiveness trial of OSCAR-S.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>65 years old)
* Scheduled to undergo an elective colorectal surgery procedure
* Ability to provide informed consent

Exclusion Criteria:

* Emergent, non-elective colorectal procedures
* Non-English Speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the implementation fidelity by the percentage of patients who complete at least two intervention touchpoints | 30 days
To determine reach by the percentage of eligible patients enrolled | 12 months
To determine effectiveness by patient satisfaction, 30-day readmission rates, mortality, and complication rates; | 30 days
To determine adoption by the percentage of providers engaging in communication with the nurse coach | 12 months
To determine maintenance fidelity by continued adherence to the protocol at 12 months | 12 months

IPD SHARING:
Plan to Share IPD: No